CLINICAL TRIAL: NCT00051584
Title: A Phase II Study of SGN-15 (cBR96 - Doxorubicin Immunoconjugate) Combined With Gemzar® Versus Single-Agent Gemzar® in Patients With Advanced Ovarian Cancer
Brief Title: Safety/Efficacy Study of SGN-15 (Antibody-Drug Conjugate) Combined With Gemcitabine in Patients With Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG015-0003; NCT00056017 (obsolete NCT alias)
Record Dates: First submitted 2003-01-13; First posted 2003-01-15 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — BR96-doxorubicin immunoconjugate; Gemcitabine

INTERVENTIONS:
Drug: SGN-15 (cBR96-Doxorubicin Immunoconjugate)
Drug: Gemzar (Gemcitabine)

SUMMARY:
This is an open-label, randomized phase II trial comparing treatment with a monoclonal antibody (mAb) drug immunoconjugate, SGN-15, administered weekly in combination with weekly Gemzar® (Gemcitabine) to treatment with Gemzar® alone. The primary objectives of this study are to determine the toxicity and safety profile of the combination of SGN-15 and Gemzar®, to estimate the clinical response rate and to estimate the duration of response of this combination therapy administered to patients with advanced ovarian cancer, compared to treatment with Gemzar® alone.

ELIGIBILITY:
Brief Overview of Inclusion Criteria:

* Patients must have pathologically confirmed ovarian cancer, which is advanced or recurrent carcinoma, who have failed at least two, but no more than three prior therapies for metastatic disease
* Patients must have > 20% Lewis-y antigen expression documented by immunohistochemistry
* LVEF > 50% by echo or MUGA
* Must be platinum resistant as defined by:

  * Progression while on initial platinum therapy or
  * Progression while on retreatment with initial platinum regimen or
  * Relapse < 6 months after initial therapy

Brief Overview of Exclusion Criteria:

* Patients who have had prior therapy with Gemzar®
* Cumulative anthracycline exposure > 300 mg/m2
* More than three prior chemotherapy regimens for ovarian cancer (Retreatment with Taxane/Platinum after initial combination is considered only one regimen)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sandler, MD, Study Director — Seagen Inc.
Locations (6):
- United States (6):
  - Arizona Cancer Center, Tucson, Arizona
  - Sharp Healthcare, San Diego, California
  - California Hematology Oncology Medical Group, Torrance, California
  - Mountain States Tumor Institute, Boise, Idaho
  - Arlington Fairfax Hematology Oncology, Arlington, Virginia
  - Virginia Mason Medical Center, Seattle, Washington